CLINICAL TRIAL: NCT02123979
Title: A Double-Blind, Placebo-Controlled, Randomized, Parallel Group Study to Assess Dopamine Receptor Modulation With Rotigotine to Enhance Opioid Analgesia Using the Oral Surgery Model of Acute Pain in Healthy Volunteers
Brief Title: Study to Assess Dopamine Receptor Modulation With Rotigotine to Enhance Morphine Analgesia in the Dental Model
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Raymond Dionne, Raymond A. Dionne, DDS, PhD Research Professor Department of Pharmacology & Toxicology Brody School of Medicine Department of Foundational Sciences School of Dental Medicine East Carolina University Greenville, NC 27834-4354, East Carolina University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-000723; 112101 668916 (Other: East Carolina University)
Record Dates: First submitted 2014-04-14; First posted 2014-04-28 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Post-op Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo patch (Placebo Comparator): Neupro® transdermal patch/placebo randomly allocated like a flip of a coin applied to your skin at the dose of 8 mg/day or a matching placebo patch after the oral surgery procedure is completed.
  Interventions: Drug: Neupro® transdermal patch/placebo
- Neupro® transdermal patch (Experimental): Neupro® transdermal patch/placebo randomly allocated like a flip of a coin applied to your skin at the dose of 8 mg/day or a matching placebo patch after the oral surgery procedure is completed.
  Interventions: Drug: Neupro® transdermal patch/placebo

INTERVENTIONS:
Drug: Neupro® transdermal patch/placebo — 8mg transdermal patch Neupro® transdermal patch/placebo
  Other Names: also known as rotigotine

SUMMARY:
Narcotics are widely used as the mainstay of pain treatment, although increasing doses are required over time as the individual becomes tolerant to their effects. This can lead to the development of dependence and abuse of these drugs. Research has identified a new way to decrease the risk of developing tolerance to narcotics, by giving at the same time a drug called rotigotine ("Neupro"). Rotigotine interferes with the body's chemical dopamine and is FDA-approved for the management of Parkinson's Disease.

The purpose of this research study is to look at side effects and pain control in healthy people after removal of wisdom teeth, which usually causes pain. It is thought that by giving the study drug rotigotine with the narcotic pain reliever, there will be pain control that will extend longer than when giving the narcotic alone.

DETAILED DESCRIPTION:
Inclusion Criteria:

* Male and female patients aged 18 and over scheduled to undergo elective oral surgery for the removal of impacted third molars
* Indicated for the removal of 3-4 third molars, at least two of which are categorized as partial-boney or full-boney impactions
* Self-report of moderate or severe pain on a categorical scale with a minimum of 5 out of 10 on the numerical rating scale following the offset of local anesthesia

Exclusion Criteria:

* History or intolerance to rotigotine
* Current or history of mental disorder or substance abuse
* Allergy or intolerance to opioids or local anesthetics
* Concurrent or recent use of agents that may confound the sedative effects of the study drug (opioids, benzodiazepines) over the previous 7 days or alcohol ingestion in the previous 24 hours
* Chronic or recent use of medications that might confound the effects of rotigotine, e.g., antihistamines, prescription or over-the-counter NSAIDs (Nonsteroidal anti-inflammatory drugs), acetaminophen, steroids, antidepressants, muscle relaxants.
* Concurrent or history of chronic diseases, e.g., diabetes, rheumatoid arthritis, liver disease, cancer, hypertension or obesity (body mass index >35).

ELIGIBILITY:
Inclusion Criteria:

* • Male and female patients aged 18 and over scheduled to undergo elective oral surgery for the removal of impacted third molars

  * Indicated for the removal of 3-4 third molars, at least two of which are categorized as partial-boney or full-boney impactions
  * Self-report of moderate or severe pain on a categorical scale with a minimum of 5 out of 10 on the numerical rating scale following the offset of local anesthesia

Exclusion Criteria:

* History or intolerance to rotigotine

  * Current or history of mental disorder or substance abuse
  * Allergy or intolerance to opioids or local anesthetics
  * Concurrent or recent use of agents that may confound the sedative effects of the study drug (opioids, benzodiazepines) over the previous 7 days or alcohol ingestion in the previous 24 hours
  * Chronic or recent use of medications that might confound the effects of rotigotine, e.g., antihistamines, prescription or over-the-counter NSAIDs, acetaminophen, steroids, antidepressants, muscle relaxants.
  * Concurrent or history of chronic diseases, e.g., diabetes, rheumatoid arthritis, liver disease, cancer, hypertension or obesity (body mass index >35).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-11 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Sum of pain intensity difference scores | up to six months
  The primary outcome measure will be the SPID (sum of pain intensity difference scores) over the 3-hour observation period for MS(morphine sulfate)+Nuepro versus MS.

SECONDARY OUTCOMES:
Analgesic tablets taken postoperatively | December 2014
  The number of analgesic tablets taken over the first 48 hours postoperatively will be compared between the two groups as a secondary measure of the ability of the D3 agonist to potentiate opioid analgesia as a surrogate indicator of reduced potential for tolerance development.

OTHER OUTCOMES:
assess pain | up 48 hours
  assess the translational potential of what has been demonstrated in the lab to human subjects experiencing painful conditions that require control with morphine. We hope to provide proof of concept for a treatment strategy that will allow opiates to maintain their effectiveness at low doses without the emergence of tolerance and other side effects, even with prolonged use.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Dionne, DDS, PhD, Principal Investigator — School of Dental Medicine, East Carolina University
Locations (1):
- School of Dental Medicine At East Carolina University, Greenville, North Carolina, United States